CLINICAL TRIAL: NCT04881539
Title: Are Natural Killer Cells Novel Mediators of the Effects of Cannabidiol on Physical Fitness, Mental Health and Well-Being, Sleep Quantity, Sleep Quantity and Immune Function?
Brief Title: CBD, Immune Function, and Neural Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Northern Colorado (Other)
Responsible Party: Principal Investigator, Laura Stewart, Professor, University of Northern Colorado
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UNColorado
Record Dates: First submitted 2021-04-21; First posted 2021-05-11 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Healthy
Keywords: CBD
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Study participants will be randomly assigned to either a CBD group or a placebo group and followed throughout the 8 week intervention period.
Who Masked: Participant, Investigator
Masking Description: A person who does not interact with the study participants will be completing the masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (CBD) (Experimental): Each group member will receive one dose of CBD daily for 8 weeks.
  Interventions: Dietary Supplement: Cannabidiol (CBD)
- Placebo (Placebo Comparator): Each group member will receive a calorie matched placebo daily for 8 weeks.
  Interventions: Dietary Supplement: Cannabidiol (CBD)

INTERVENTIONS:
Dietary Supplement: Cannabidiol (CBD) — This group will receive an oral dose of CBD (Six Degrees Wellness).

SUMMARY:
Chronic inflammation, which is defined as a persistent, low-grade inflammatory response within the body, is associated with many of the negative health conditions which are prevalent in our society today. It is most well-known for its role in the progression of diseases including obesity, metabolic syndrome, cancer, cardiovascular disease, and diabetes. Chronic inflammation is also linked to many of the underlying factors associated with disease development including perturbations in sleep, and mental health status such as depression, anxiety, fatigue, and quality of life. Natural killer cells, commonly referred to as NK cells, are a subset of white blood cells that play an important role in the coordination of inflammation in the body.

Although many interventions aimed at controlling chronic inflammation and enhancing NK cell number and activity have been explored, relatively few have been administered without significant barriers. Cannabidiol (CBD), a non-psychoactive hemp derivative, is a potential, attractive therapeutic target. However, there is very little information in humans that addresses the potential of CBD to improve your health and immune function.

The overall goal of this study is to explore the effects of 8-weeks of CBD supplementation on mental and physical health, sleep measures, and NK cell number and cytotoxic function. Specific Aim 1. Explore the effect of 8-weeks of CBD administration on sleep measures as well as measures of mental and physical health in conjunction with measurements of NK cell number and function.

DETAILED DESCRIPTION:
In this double-blind investigation, participants will undergo 8 total visits separated by an 8-week intervention period. One week prior to the intervention period, participants will complete a blood draw, body composition analysis, aerobic and anaerobic fitness analysis, maximal strength testing, and physical activity and sleep quantity and quality analyses. These tests will be completed again following the 8-week intervention period. Following the first 4 visits, participants will be randomly assigned 1 of 2 groups: CBD (50mg/day) or calorie matched placebo. Participants will then complete the 8-week intervention period. Additionally, during week 4 of the 8-week intervention period (intervention midpoint), participants will complete a blood draw, one full week of physical activity and sleep actigraphy, surveys on mental health and wellbeing, and prevalence of sickness and illness

ELIGIBILITY:
Inclusion Criteria:

* Participants must be within 18 and 50 years of age
* Abstained from cannabis (either THC and/or CBD) for the past 6 weeks
* Have a BMI of 29.9 or below
* Completes at least 150 minutes of moderate to vigorous physical activity per week.
* Able and willing to commit to an 8-week intervention schedule

Exclusion Criteria:

* Significant cardiovascular disorders including but not limited to serious arrhythmias, cardiomyopathy, congestive heart failure, stroke, or transient ischemic attacks, peripheral vascular disease with intermittent claudication, acute, chronic or recurrent thrombophlebitis.
* Diagnosed neurological disorders including but not limited to brain tumors, brain injuries, Alzheimer's Disease, Parkinson's Disease, multiple sclerosis, epilepsy, and seizures.
* Regular use of drugs that significantly alter brain activity such as selective serotonin reuptake inhibitors, benzodiazepines, and others used to treat anxiety, panic, stress, sleep disorders, or increases the risk of sedation and drowsiness.
* Head trauma with loss of consciousness for more than 30 mins.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Individuals will be asked to self select their biological sex.
Enrollment: 50 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Natural Killer Cell Number | 8 Weeks
  We will use a flow cytometry to evaluate natural killer cell number and function before and after the intervention.
Natural Killer Cell Number and Function | 8 Weeks
  We will use a flow cytometry to evaluate natural killer cell number and function before and after the intervention.
Physical Activity | 8 Weeks
  We will use a Fitbit to track physical activity before and after the intervention.
Sleep | 8 Weeks
  We will use a Fitbit Sleep Tracker before and after the intervention.
Immune Biomarker (C-Reactive Protein (CRP)) | 8 Weeks
  We will measure serum CRP in pre and post intervention samples.
Immune Biomarker (Interleukin 6 (IL-6)) | 8 Weeks
  We will measure serum Il-6 in pre and post intervention samples.
Neural Health Biomarker (Brain Derived Neurotrophic Factor (BDNF)) | 8 Weeks
  We will measure circulating BDNF in pre and post intervention samples.
NK Cell Function | 8 Weeks
  We will use a flow cytometry to evaluate natural killer cell number and function before and after the intervention.

SECONDARY OUTCOMES:
Body Composition | 8 Weeks
  We will use the Bod Pod before and after the intervention to evaluate body composition.
Anaerobic Fitness | 8 Weeks
  We will test subject ability to perform a Wingate Power Test before and after the intervention.
Cognitive Function Questionnaire | 8 Weeks
  We will evaluate cognitive function with the PROMIS SF v. 2.0 Abilities Questionnaire before and after the intervention. A higher score suggests higher cognitive ability.
Anxiety Questionnaire | 8 Weeks
  We will use the General Anxiety Disorder -7 Questionnaire before and after the intervention. The higher the score suggests higher levels of anxiety.
Sleep Evaluation Questionnaire | 8 Weeks
  We will use the Leeds Sleep Evaluation Questionnaire before and after the intervention. Lower scores generally suggest better sleep.
Depression Questionnaire | 8 Weeks
  We will use the Beck Depression Inventory before and after the intervention period. A higher score on this survey suggests the presence of more depression.
Strength Assessment | 8 Weeks
  All subjects will complete a 1 repetition or 8 repetition max back squat test before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Stewart, PhD, Principal Investigator — University of Northern Colorado
Locations (1):
- University Of Northern Colorado, Greeley, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification will be available
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately after publication date for 3 years.
Access Criteria: Proposals should be directed to laura.stewart@unco.edu